CLINICAL TRIAL: NCT06943625
Title: Combined Effects of Green Light and Transcranial Direct Current Stimulation on Migraine Intensity and Frequency in Migraine Patients.
Brief Title: Combined Effects of Green Light and Transcranial Direct Current Stimulation in Migraine Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC02167 Sufia Umar
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: migraine; neuromodulation; brain stimulation
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation; Green Light; Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): tDCS will applied to the participants of this group along with medication advised
  Interventions: Other: tDCS; Other: medicine
- Group 2 (Active Comparator): Green light exposure will be provided to the participants of this group along with the medications advised.
  Interventions: Other: Green light; Other: medicine
- Group 3 (Experimental): tDCS and green light will be provided to the participants of this group along with the medications advised
  Interventions: Other: tDCS; Other: Green light; Other: medicine
- Group 4 (Active Comparator): Only advised medication will be utilized by the participants in this group
  Interventions: Other: medicine

INTERVENTIONS:
Other: tDCS — Transcranial direct current stimulation protocol involves 20 minutes of anodal stimulation, with the anodal electrode placed over the motor cortex (primary motor area), and cathodal stimulation applied to the contralateral supraorbital area.
  The intensity of the current will be set to 1.5 mA, with the current density ranging from approximately 0.03 to 0.06 mA, with the electrode measuring of 5x7cm. To ensure a gradual and comfortable experience for participants, the current will ramp up and down over 30 seconds at the beginning and end of each session. Each stimulation session will last for 20 minutes, with participants undergoing five sessions per week. The entire intervention protocol will be carried out over a period of four weeks
  Arms: Group 1; Group 3
Other: Green light — Green light exposure will be administered using light with a wavelength of about 520 nm. The sessions will take place in a dimly lit room to minimize external light interference and enhance the therapeutic effect of the green light. Each exposure session will last for 2 hours, with participants receiving 3 to 5 sessions per week. The light intensity will be set to 100 lux, a level that is both safe and effective for migraine treatment. The entire intervention protocol will span over four weeks to allow for sufficient evaluation of the effects. During each session, participants will be seated comfortably in a chair to ensure they are relaxed and able to tolerate light exposure without discomfort.
  Arms: Group 2; Group 3
Other: medicine — Advised medicine by the medical doctors will be utilized by the participants of the study

SUMMARY:
According to the Global Burden of Disease (GBD) study, headache disorders are among the most prevalent and disabling conditions worldwide, with estimated 1-year prevalence of migraine (22.5%) in Pakistan, considerably higher than the global 1-year prevalence of 15%.

The treatment options comprise such as lifestyle modifications, behavioral therapy, medication such as nonsteroidal anti-inflammatory drugs (NSAIDs), beta blockers, calcium channel blockers, antiepileptic drugs or antibodies against calcitonin gene-related peptide (CGRP) or its receptor, and neuromodulation.

One of the non-invasive neuromodulation technique is used in migraine patients .i.e., transcranial direct current stimulation (tDCS), tDCS is a promising method for migraine treatment delivering a low-intensity current through the scalp by means of electrodes to modulate the state of polarization of the cerebral cortex; depending on the polarity of the electrical stimulation, tDCS can be either anodal(excitatory) or cathodal(inhibitory). Neuromodulation by tDCS is thought to follow Hebbian Theory ("neurons that fire together, wire together"). If presynaptic and postsynaptic neurons are both active, the result is synaptic strengthening; if one or both are inactive, no change occurs. The literature reported significant reduction in migraine days when applying tDCS to the occipital cortex, primary motor cortex, or the dorsolateral prefrontal cortex. The advantages of tDCS treatment are its relatively low cost compared to other neurostimulator methods, safety and generally mild side effects.

DETAILED DESCRIPTION:
Migraine is a common and debilitating neurological disorder, defined as "an episodic headache associated with certain features, such as sensitivity to light, sound, or movement", classified by headache frequency, with chronic migraine (CM), defined as 15 or more headache days a month for three or more months while episodic migraine (EM), is defined as occurring on fewer than 15 headache days per month.

It is also known as a common relapsing headache disease with a huge socioeconomic burden, characterized by a headache lasting 4 - 72 hours when untreated, which tends to be unilateral, pulsating, and of moderate to severe pain intensity.

According to the Global Burden of Disease (GBD) study, headache disorders are among the most prevalent and disabling conditions worldwide, with estimated 1-year prevalence of migraine (22.5%) in Pakistan, considerably higher than the global 1-year prevalence of 15%.

In the international classification of headache disorders 3rd Edition (ICHD-3), migraines may be diagnosed with aura or without aura. Migraine with aura is a complex neurological manifesting clinically as visual, somatosensory, speech or motor symptoms that precedes the headache phase. Migraine without aura is a recurrent headache disorder with specific features like unilateral, pulsating pain, nausea, and light/sound sensitivity, lasting between 4 and 72 hours.

The Graham and Wolff proposed the vascular theory for migraines, which stated that the serotonin released from the platelets in blood vessels to be the causal molecule. Because serotonin has constrictive effects on blood vessels, local cerebral blood flow is decreased, and this was thought to cause the auras that occur in migraines. After the reuptake or metabolism of this serotonin, the constricted blood vessels dilate, inducing the pain of the migraine headache.

The primary cause of migraines is the activation of the cervical complex of the trigeminal nucleus and trigeminal nerve. This activation of the trigeminal nerve results in neurogenic inflammation, including CGRP release from the C-fibers of the trigeminal ganglion and peripheral trigeminal nerve terminal. CGRP receptors are located in larger neurons and thicker fibers, which correspond to the Aδ-fibers of the trigeminal nerve. A δ-fibers are myelinated nociceptive nerves; thus, stimulation of Aδ-fiber CGRP receptors causes sharp severe headaches. The activation of the trigeminovascular system, mostly pertaining to the peripheral nervous system, is the key event of migraine pain generation.

The treatment options comprise such as lifestyle modifications, behavioral therapy, medication such as nonsteroidal anti-inflammatory drugs (NSAIDs), beta blockers, calcium channel blockers, antiepileptic drugs or antibodies against calcitonin gene-related peptide (CGRP) or its receptor, and neuromodulation. Neuromodulation can be defined as an intervention that potentiates or inhibits the transmission of a nerve impulse but is not the actual means of transmission itself.

One of the non-invasive neuromodulation technique is used in migraine patients .i.e., transcranial direct current stimulation (tDCS), tDCS is a promising method for migraine treatment delivering a low-intensity current through the scalp by means of electrodes to modulate the state of polarization of the cerebral cortex; depending on the polarity of the electrical stimulation, tDCS can be either anodal(excitatory) or cathodal(inhibitory). Neuromodulation by tDCS is thought to follow Hebbian Theory ("neurons that fire together, wire together"). If presynaptic and postsynaptic neurons are both active, the result is synaptic strengthening; if one or both are inactive, no change occurs. The literature reported significant reduction in migraine days when applying tDCS to the occipital cortex, primary motor cortex, or the dorsolateral prefrontal cortex. The advantages of tDCS treatment are its relatively low cost compared to other neuro-stimulation methods, safety and generally mild side effects.

Reports suggested that exposure to lights of different wavelengths can affect nociception in rodents. For example, exposure to a green light emitting diode (GLED) resulted in anti-nociception in naïve rats and anti-hyperalgesia in rats with neuropathic pain that was dependent on engagement of the visual system. Also exploratory studies demonstrated that isolated exposure to green light may reduce the intensity and duration of migraine attacks.

The rationale for this study is to evaluate whether combining tDCS with green light exposure provides synergistic benefits in reducing migraine frequency, intensity, and improving the overall quality of life for patients suffering from migraine. This dual approach may enhance therapeutic outcomes by targeting both the neural mechanisms underlying migraine attacks through neuromodulation (tDCS) and alleviating visual discomfort via green light.

The proposed study seeks to address a gap in current migraine treatment by exploring the potential of a non-pharmacological, combinatory intervention that could offer a more effective, lasting solution for migraine management. Given the growing interest in non-pharmacological treatments for migraine and the promise of both tDCS and green light exposure, this research will hold significant potential for advancing migraine care and providing new treatment options for patients who prefer or require alternatives to conventional medications.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine or chronic migraine according to the International Headache Society
* An average headache pain intensity of migraine episodes of ≥5 at numeric pain scale (NPS) over the 4 weeks prior to enrolling in the study

Exclusion Criteria:

* Mental illness
* Photophobic individual
* Presence of shunt and/or implant at the cranial region
* Brain tumors
* Wound at skull

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Structured Headache Diary Data | 4 week
  Structured Headache Diary Data for frequency of migraine
Numeric Pain Scale | 4 week
  Numeric Pain Scale (NPS) for intensity of migraine, is a simple 0-10 tool for measuring pain intensity, where 0 is "no pain" and 10 is "worst pain

SECONDARY OUTCOMES:
Multidimensional Pain Inventory | 4 week
  Multidimensional Pain Inventory (MPI) for migraine impact, is scored by summing responses to specific items (rated 0-6) for various subscales, then calculating a mean score (e.g., (Q1+Q7+Q12)/3 for Pain Severity), providing 12 distinct scores across Pain Impact, Significant Other Responses, and Activity levels, helping clinicians understand pain's breadth, not just severity, with higher scores generally indicating greater impact or distress, though some scales (like Activity) use higher scores for more function.
Migraine-Specific Quality of Life Survey | 4 week
  Migraine-Specific Quality of Life Survey (MSQ 2.1) for quality of life, involves rating 14 items on a 6-point scale (1=All the time, 6=None of the time) across three domains (Role-Restrictive, Role-Preventive, Emotional Function), summing item scores, and then rescaling them to a 0-100 scale where higher scores mean better quality of life, reflecting how migraines impact daily activities, work, and feelings over the past four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moisset X, Pereira B, Ciampi de Andrade D, Fontaine D, Lanteri-Minet M, Mawet J. Neuromodulation techniques for acute and preventive migraine treatment: a systematic review and meta-analysis of randomized controlled trials. J Headache Pain. 2020 Dec 10;21(1):142. doi: 10.1186/s10194-020-01204-4. PMID 33302882
- [Background] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119